CLINICAL TRIAL: NCT06819748
Title: Efficacy and Safety of Cocktail of Ropivacaine,sodium Bicarbonate and Dexamethasone for Incision Local Infiltration Analgesia in Patients Undergoing Ambulatory Laparoscopic Cholecystectomy:A Prospective Randomized Control Trial
Brief Title: Efficacy and Safety of Cocktail of Ropivacaine for Local Infiltration Analgesia in Patients Undergoing Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Xia Zhiying, resident physician, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20247411
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Cholecystectomy, Laparoscopic; Ambulatory Surgical Procedures; Multimodal Analgesia
MeSH Terms: interventions — Dexamethasone; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A group (Experimental): Drug:cocktail of 0.5% ropivacaine ,5%sodium bicarbonate and 10mg dexamethasone
  Interventions: Drug: The cocktail of 0.5% ropivacaine ,5%sodium bicarbonate and 10 mg dexamethasone
- B group (Active Comparator): Drug: 0.5%ropivacaine
  Interventions: Drug: 0.5% ropivacaine

INTERVENTIONS:
Drug: The cocktail of 0.5% ropivacaine ,5%sodium bicarbonate and 10 mg dexamethasone — The patient receive the cocktail of 0.5% ropivacaine ,5%sodium bicarbonate and 10 mg dexamethasone as incision local anesthesia at the end of surgery
  Other Names: 0.5% ropivacaine; The cocktail of ropivacaine
  Arms: A group
Drug: 0.5% ropivacaine — The patient receive 0.5% ropivacaine as incision local anesthesia at the end of surgery
  Arms: B group

SUMMARY:
The goal of this clinical trial is to learn if the use of cocktail of ropivacaine,sodium bicarbonate and dexamethasone for incision local infiltration analgesia in patients undergoing ambulatory laparoscopic cholecystectomy is safe and effective. The main questions it aims to answer are:

Does the cocktail lower the The incidence of moderate to severe pain during movement stages within six hours after surgery.

Researchers will compare the cocktail to ropivacaine for incision local infiltration analgesia to see if the cocktail works to moderate the postoperative pain of ambulatory laparoscopic cholecystectomy patients.

Participants will:

Receive the cocktail or ropivacaine for incision local infiltration analgesia at the end of the surgery.

Answer the questions about postsurgical pain at rest or during motion(using a Numeric Rating Scale (NRS) of 0 to 10. Pain measurements were performed at 2, 6, 12, 24 hours,3,7,30 days and 3 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing daytime laparoscopic cholecystectomy in Sichuan Provincial People's hospital ② Age: 18-70 years

  * American society of Anesthesiologists physical status classification system I-II ④ 18 kg/㎡≤ BMI ≤ 30 kg/㎡ ⑤ No communication barriers, able to understand the research process and the use of pain scale.

    * Signed informed consent

Exclusion Criteria:

* Drug allergy related to this study

  * History of chronic pain, long-term use of analgesic drugs (equivalent to ≥ 10mg oxycodone per day), alcohol abuse, gastrointestinal bleeding or perforation after application of non steroidal anti-inflammatory drugs

    * Patients with ischemic heart disease, peripheral arterial vascular or cerebrovascular disease, or patients with pulmonary heart disease, active peptic ulcer or gastrointestinal bleeding, or patients with inflammatory bowel disease

      * Patients taking monoamine oxidase inhibitors or within 2 weeks after discontinuation ⑤ Preoperative pain score (NRS ) was greater than or equal to 4 points ⑥ Participated in other clinical studies within three months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of moderate to severe pain（Numerical Rating Scale) during movement stages within six hours after surgery | 2, 6, 12, 24 hours,3,7,30 days and 3 months postoperatively
  The result is quantified continuously in a scale from 0 (No pain) to 10 (Worst pain imaginable) points. Acute pain is labeled of a value ≥4 points.

SECONDARY OUTCOMES:
Number of Participants With Opioid Administration | 2, 6, 12, 24 hours postoperatively
  The administration of opioids in the first two hours of postoperative for necessary reasons (pain ≥4 points) is recorded by the physician in charge.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Fan, M.D/PhD, Principal Investigator — Sichuan Provincial People's Hospital
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided